CLINICAL TRIAL: NCT03731754
Title: "Cross" Closure for Reconstructing the Perineal Wound of Abdominoperineal Resection in Rectal and Anal Cancer Patients: a Multi-center, Randomized, Open-Label, Positive, Parallel Controlled Clinical Trial
Brief Title: "Cross" Closure for Reconstructing the Perineal Wound of Abdominoperineal Resection
Acronym: CCRPWAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); First Affiliated Hospital of Jinan University (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); Southern Medical University, China (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Guangzhou First People's Hospital (Other); Affiliated Hospital of Guangdong Medical University (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Meizhou People's Hospital (Other); Jieyang People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCRPWAR
Record Dates: First submitted 2018-10-26; First posted 2018-11-06 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-10

CONDITIONS: Rectal Cancer; Anal Canal Cancer
Keywords: Traditional closure; "Cross" closure; Rectal cancer; Anal canal cancer; Abdominoperineal resection
MeSH Terms: conditions — Rectal Neoplasms; Anal Canal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Closure (Active Comparator): Patients receive primary closure discontinuously for reconstruction of APR perineal wound
  Interventions: Procedure: Traditional Closure
- "Cross" Closure (Experimental): Patients receive "cross" closure for reconstruction of APR perineal wound
  Interventions: Procedure: "Cross" closure

INTERVENTIONS:
Procedure: Traditional Closure — Primary closure discontinuously the perineal wound of APR
  Arms: Traditional Closure
Procedure: "Cross" closure — Two triangles of skin in the horizontal direction are excised to enlarge the skin incision, and the tumor resected. Then circumferential subcuticular suture of wound, and with tightening of the circumferential suture, the wound resembles a cross.
  Arms: "Cross" Closure

SUMMARY:
How to reduce the complications of perineal wound after abdominoperineal resection (APR) has always been a hot topic in the medical field.To reduce the complications of perineal wound and the primary healing of perineal wound must meet the two principles of "unobstructed drainage" and " reduced tension closure".This concept is similar to the concepts of closure of enterostomy in rectal cancer patients. It was reported that use of cross-stitch closure can significantly reduce complications of closure of enterostomy. So the investigator ever used the "cross" closure to reconstruct the perineal wound of APR, which was really decrease the complications of perineal wound. However, more clinical trails was needed to confirm the conclusion.

DETAILED DESCRIPTION:
Perineal wound problems after abdominoperineal resection (APR) for rectal cancer is reported in up to 25%～66% of patients,if the perineum does not heal primarily, the secondary wound healing may prolong hospital stay, may necessitate surgical reintervention, and often requires intensive wound care for several months. Great efforts have been taken to reduce the complications of perineal wound of APR, but the incidence of the perineal wound complications are not effectively decreased.

It was reported that one of the most important factors to determine the primary healing of perineal wound is whether the anterior sacral drainage and perineal stump drainage are sufficient and effective or not, which is similar to the concept of closure of enterostomy.

Previously, it was reported that "cross" closure is an effective method of skin closure for stoma reversal, which allows increased surgical exposure, reduces suture, smooth drainage, aesthetic healing simplifies wound care, and gives a neat cosmetic result.

Therefore, because of the success use of "cross" closure in stoma reversal to reduce the complications of perineal wound, the investigator used the "cross" closure to reconstruct the perineal wound of APR, and it really can decrease the complications of perineal wound. However, more clinical trails are needed to confirm the conclusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years old;
2. ECOG performance status: 0-2;
3. Histologically confirmed rectal cancer or anal canal cancer;
4. Completely resected the primary tumor;
5. No evidence of distant metastasis;
6. Tolerable general anesthesia;
7. Total radiation dose of 45-50 Gy needed if the patient needs to receive routine segmental radiotherapy;
8. Provision of written informed consent.

Exclusion Criteria:

1. Emergency surgery required when the patients combined with acute ileus, perforation and hemorrhage;
2. Extralevator abdominoperineal resection needed;
3. American Society of Anesthesiologists (ASA) IV or V;
4. Combined with other tumors;
5. Severe mental illness;

(7)Serious cardiovascular disease, uncontrolled infections, or other serious uncontrolled concomitant disease; (8)Expectation of lateral lymph node dissection preoperatively

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Estimated)
Dates: Start 2018-11-20 (Estimated); Primary Completion 2020-11-20 (Estimated); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
Complication rate of perineal wound | Within 30 days after operation
  the complications of perineal wound are include wound infection, wound effusion, wound liquefaction, wound dehiscence, seroma or hematoma ,delayed wound healing, presacral or perineal abscess, perineal or pelvic floor hernia

SECONDARY OUTCOMES:
Primary wound healing rate | Within 30 days after operation
  the Primary wound healing rate within 30 days after operation
CTCAE grade for complications of perineal wound | Within 30 days after surgery
  the CTCAE grade for complications of perineal wound within 30 days after surgery
The incidence of each complication of perineal wound | Within 30 days after surgery
  The incidence of each complication of perineal wound within 30 days after surgery
The rate of reoperation | Within 30 days after surgery
  The rate of reoperation within 30 days after surgery
The volumes of presacral drainage | Within 3, 5, 7 days after surgery
  The volumes of presacral drainage within 3, 5, 7 days after surgery
The volumes of presacral residual cavity hydrops | 3 and 7 days postoperatively
  The volumes of presacral residual cavity hydrops within 3 and 7 days postoperatively
The times of dressing change of perineal wound | Within 3, 5, 7 days after surgery
  The times of dressing change of perineal wound within 3, 5, 7 days after surgery
Removal time of presacral drainage tube | Within 30 days after surgery
  Removal time of presacral drainage tube within 30 days after surgery
Scar scores for perineal wound and evaluation of patients' overall satisfaction | Within 30 days after surgery
  Scar scores for perineal wound and evaluation of patients' overall satisfaction within 30 days after surgery
Hospital stay after surgery | Within 30 days after surgery
  Hospital stay after surgery within 30 days after surgery
The operation time | Intraoperatively
  The operation time

CONTACTS AND LOCATIONS:
Overall Officials: Lei Wang, MD, PhD, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University